CLINICAL TRIAL: NCT05887921
Title: Inguinal Lymphadenectomy for Penile Cancer: an Interim Report From a Prospective Randomized Clinical Trial Comparing Open vs. Video-endoscopic Approach
Brief Title: Inguinal Lymphadenectomy for Penile Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Mirko Preto, MD, PhD, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00025/2020
Record Dates: First submitted 2022-12-29; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Penile Cancer; Lymph Node Metastasis; Sentinel Lymph Node; Surgical Complication
MeSH Terms: conditions — Penile Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: Surgical, observational, prospective, monocentric study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open inguinal Lymphadenectomy (Active Comparator): - Groin 1: open lymphadenectomy performed by a surgical team with extensive experience in traditional surgery
  Interventions: Procedure: Inguinal Lymphadenectomy
- Laparoscopic inguinal Lymphadenectomy (Active Comparator): Groin 2: laparoscopic lymphadenectomy performed by a surgical team with extensive experience in minimally invasive surgery
  Interventions: Procedure: Inguinal Lymphadenectomy

INTERVENTIONS:
Procedure: Inguinal Lymphadenectomy — arm A: open lymphadenectomy performed by a surgical team with extensive experience in traditional surgery arm B: laparoscopic lymphadenectomy performed by a surgical team with extensive experience in minimally invasive surgery

SUMMARY:
The aim of the present study is to prospectively compare oncological and functional results of penile radical inguinal lymphadenectomy performed with an open versus videolaparoscopic technique.

The main questions it aims to answer are: evaluated the oncological and functional results of inguinal lymphadenectomy performed with minimally invasive techniques using videolaparoscopic instruments vs open inguinal lymphadenectomy according to the standard technique.

Participants will undergo treatment of the primary lesion and contextual inguinal lymphadenectomy:

* Groin 1: open lymphadenectomy performed by a surgical team with extensive experience in traditional surgery
* Groin 2: laparoscopic lymphadenectomy performed by a surgical team with extensive experience in minimally invasive surgery. The results of these procedures will be prospectively collected and compared.

DETAILED DESCRIPTION:
Penile cancer represents, to date, a rare oncological pathology (1/100000 males in Europe). However, in tertiary reference centres, such as the SCU Urologia (Prof. P.

Gontero), the number of patients sent for this pathology is increasing. Although for the main lesion (T) there are now consolidated standards of care, increasingly aimed at a conservative "sexual sparing" approach where oncologically possible, the management of loco-regional lymph nodes is still not completely standardized. The European Guidelines (EAU) recommend bilateral inguinal radical lymphadenectomy for cN1/N2 (palpable lymph nodes mono/bilaterally, but not fixed) or high-risk tumour (> T1G2). Lymph node management is the factor that most influences patient survival. For this reason, this must be entrusted to highly specialized centres. Some recent trials have shown that bilateral inguinal lymphadenectomy has a statistically significant superiority to radiotherapy and clinical surveillance in cN1/N2 patients. Despite this, inguinal lymphadenectomy has an important incidence of morbidity (up to 50% of cases) which often wrongly limits its indications. Main complications are: Lymphocele

* Prolonged lymphatic drainage
* Skin necrosis
* Dehiscence of the surgical wound
* Edema of lower limbs and genitals Only few studies have recently evaluated the oncological and functional results of inguinal lymphadenectomy performed with minimally invasive techniques using videolaparoscopic instruments. First results seem to support minimally invasive approach, that appears to have comparable oncological results and less post-operative morbidity.

However, evidences are still extremely limited, and no high-grade recommendations can be made. The aim of the present study is to prospectively compare oncological and functional results of penile radical inguinal lymphadenectomy performed with an open versus videolaparoscopic technique.

20 patients with indication for inguinal lymphadenectomy (according to EAU 2019 Guidelines - in case of primary lesion > pT1G2 or in case of lymph node disease cN1/N2) will be enrolled. Each patient will undergo treatment of the primary lesion and contextual inguinal lymphadenectomy. The procedure will be performed in this way:

* Groin 1: open lymphadenectomy performed by a surgical team with extensive experience in traditional surgery
* Groin 2: laparoscopic lymphadenectomy performed by a surgical team with extensive experience in minimally invasive surgery The results of these procedures will be prospectively collected and compared. The main outcome will be the percentage of postoperative complications (lymphocele, prolonged lymph drainage, necrosis of the skin, dehiscence of the surgical wound, edema of lower limb, emergency admission from the ED, re-intervention/surgical revision).

Complications will be classified according to the international Clavien-Dindo classification. Additionally, secondary outcomes (number of lymph nodes, number of positive lymph nodes, surgical time) will be evaluated. After the operation, patients will attend a 24-month follow-up program, as reported in the flow chart, functional results and patient satisfaction will be evaluated during the visits.

The categorical variables will be described using frequency and percentage, and the continuous variables will be described using median and interquartile range (IQR) value.

Differences between groups will be assessed by the Student independent t test or the Mann-Whitney U test on the basis of their normal or not-normal distribution, respectively (normality of variables' distribution will be tested by the Kolmogorov-Smirnov test).

ELIGIBILITY:
Inclusion Criteria:

Age of patients [45-80], CCI ≤ 3. Penile tumour with inguinal lymphadenectomy indication, according to EAU 2019 guidelines. Written informed consent.

Exclusion Criteria:

Age of patients> 80, CCI ≥ 3. Patients with lymphatic disorders of lower limbs. Patients with previous inguinal surgery/radiotherapy. Previous or concomitant diagnosis of other tumours.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with a diagnosis of penile cancer
Enrollment: 14 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Surgical outcomes of lymph drainage (ml) | 24 months
  Stratification of complications according to the international classification of Clavien-Dindo.

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U. Città della Salute e della Scienza di Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: No
All the data are anonymous and cannot be reconducted to patients if the legend is not available.
  this legend is owned only by the principal investigator

REFERENCES:
- [Derived] Falcone M, Gul M, Peretti F, Preto M, Cirigliano L, Scavone M, Sedigh O, Oderda M, Gontero P. Inguinal Lymphadenectomy for Penile Cancer: An Interim Report from a Trial Comparing Open Versus Videoendoscopic Surgery Using a Within-patient Design. Eur Urol Open Sci. 2024 Mar 21;63:31-37. doi: 10.1016/j.euros.2024.02.007. eCollection 2024 May. PMID 38558767

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT05887921/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT05887921/ICF_001.pdf